CLINICAL TRIAL: NCT05377450
Title: Prospective Randomized Study of Cementless Versus Cemented Unicompartmental Knee Arthroplasty (UKA)
Brief Title: Prospective Randomized Study of Cementless vs Cemented UKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JIS Research Institute (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-Engage PKA
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cemented Engage Partial Knee (Active Comparator): Engage partial knee implanted with bone cement for fixation.
  Interventions: Device: Engage Partial Knee
- Cementless Engage Partial Knee (Active Comparator): Engage partial knee implanted with cementless fixation.
  Interventions: Device: Engage Partial Knee

INTERVENTIONS:
Device: Engage Partial Knee — Unicompartmental knee arthroplasty utilizing the Engage Partial Knee system with bone cement.
  Arms: Cemented Engage Partial Knee
Device: Engage Partial Knee — Unicompartmental knee arthroplasty utilizing the Engage Partial Knee system without bone cement.
  Arms: Cementless Engage Partial Knee

SUMMARY:
To evaluate the non-inferiority of the cementless Engage Partial Knee System compared to cemented Engage Partial knee System.

DETAILED DESCRIPTION:
Medial unicompartmental knee arthroplasty has demonstrated outstanding success in the treatment of anteromedial osteoarthritis of the knee. Most UKA implants in the US market require cemented fixation, and there can be specific complications related to cement such as aseptic loosening between the bone-cement and/or cement-implant interface along with loose cement causing third-body wear of the remaining normal articular cartilage. Cementless devices offer a durable long-term fixation method with no risk of loose cement causing secondary damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-operative Knee Society Assessment Score of <70
* Patients undergoing primary partial knee arthroplasty as unilateral arthroplasty or bilateral arthroplasty, simultaneously or otherwise
* Patients diagnosed with osteoarthritis (Kellgren Lawrence Grade IV) or avascular necrosis limited to the medial compartment of the operative knee joint
* Male or female patients who are at least 21 years of age at the time of surgery
* Patients with full thickness cartilage loss, with or without bone loss in the medial compartment
* Patients with functionally intact ACL and PCL
* Patients who need to obtain relief of pain and/or improved function in their knee
* Patients with fixed flexion deformity < 15°
* Patients who are able to follow post operative care instructions
* Patients who are willing and able to return for scheduled follow-up evaluations
* Patients in which natural alignment can be restored
* Patients with BMI < 40
* Patients who have completed a valid, IRB approved Informed Consent Form

Exclusion Criteria:

* Patients with a pre-operative Knee Society Assessment Score of ≥ 70
* Patients in which the device would be used to revise a failed prosthesis
* Patients who are less than 21 years of age at the time of surgery
* Disease or damage to the lateral part of the knee that in the investigator's opinion contraindicates a partial knee replacement
* Patients diagnosed with rheumatoid arthritis or other forms of inflammatory joint disease
* Patients diagnosed with a failed upper tibial osteotomy in the operative knee
* Patients diagnosed with post-traumatic arthritis after tibial plateau fracture
* Patients who have had a patellectomy
* Patients with a flexion deformity > 15°
* Patients with a fixed varus deformity > 15°
* Patients who have rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Patients with a fused knee on operative side
* Patients who have active or suspected infection, local or systemic that, in the opinion of the investigator, may put patients at undue risk.
* Patient with pre-existing condition(s) that may interfere with the survival of the implant or their outcomes, including: Sickle Cell Anemia, Lower extremity muscular atrophy, Neuromuscular disease, Vascular insufficiency, Metabolic Disorders which impair bone formation, Paget's Disease, Charcot's Disease, Osteomalacia, Osteoporosis, Osteopenia.
* Patients with clinical conditions that may limit follow-up (in the opinion of the investigator) including: Immuno-compromised conditions (i.e. HIV), Hepatitis, Tuberculosis, Neoplastic disease such as cancer of the prostate, lung, stomach, cervix, etc.
* Chronic renal failure
* Organ transplant (i.e., heart, liver, lung, etc.) recipients
* Known disease process that in the opinion of the investigator may limit long term (4 year) follow up (i.e., multiple sclerosis, leukemia, lymphoma, etc.)
* Patients diagnosed with Parkinson's or Alzheimer's Disease
* Patients who have had an above-knee amputation in the contralateral leg Instability or deformity of the ligaments and/or surrounding soft tissue, which would preclude stability of the prostheses
* Patients with a known metal allergy
* Prisoners or, individuals who are known to be abusing drugs or alcohol or are mentally incompetent
* Patients who have received systemic steroids within the past 6 months or steroid injection into the affected knee within the previous 6 weeks prior to enrollment
* Patients taking immunosuppressives
* Patients who are pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study
* Patients with severe valgus or varus knees (valgus or varus angulation of more than 20°) where collateral ligament, iliotibial band, or popliteal release is required
* Patients who refuse to sign the IRB approved Informed Consent Form
* Participation in an interventional clinical research study procedure, other than a bilateral knee arthroplasty in this study, within the past 12 months
* Patients with a history of osteomyelitis or sepsis of the index knee
* Patients who require patellar resurfacing
* Patients who are not skeletally mature
* Patients who have had a total hip replacement procedure <18 months prior to entering the study
* Patients who have had a contralateral non-study knee replacement procedure <18 months prior to entering the study
* Patients who are found intraoperatively to have inadequate bone stock or other conditions that contraindicate a partial knee replacement
* Patients who have a higher risk of falling
* Patients who are smokers or a history of smoking in the past 12 months
* Patients with alcoholism or drug addiction
* Tumors of the supporting bone structures
* Patients who have a permanent valgus or varus deformity including tibia vara deformity
* Patients with BMI ≥ 40
* Patients 80 years of age or older
* Patients who have undergone same-day or staged bi-lateral partial knee replacement
* Patients who may have an allergic reaction to the device materials or bone cement

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
KOOS JR Score | 2 Years
  KOOS JR is a survey evaluating knee health for individuals following joint replacement by evaluating stiffness, pain, function, and activities of daily living.

SECONDARY OUTCOMES:
Pain Score | 6 weeks; 3, 6, 9, 12 and 24 months
  Patient rated operative knee pain on a Likert pain score of 0-10.
Range of Motion | 6 weeks; 3, 6, 9, 12 and 24 months
  Patient's range of motion is a measurement of the operated knee's extension and flexion.
KOOS JR Score | 6 weeks; 3, 6, 9, and 12 months
  KOOS JR is a survey evaluating knee health for individuals following joint replacement by evaluating stiffness, pain, function, and activities of daily living.
Implant Survivorship | 2 Year
  Implant survivorship will be determined using revision surgery on the operated knee as implant failure.

CONTACTS AND LOCATIONS:
Overall Officials: David A Crawford, MD, Principal Investigator — JIS Research Institute
Locations (1):
- JIS Research Institute, New Albany, Ohio, United States

IPD SHARING:
Plan to Share IPD: No